CLINICAL TRIAL: NCT01506791
Title: Randomized, Open-Label, 2-Way Crossover, Bioequivalence Study of Desloratadine and Pseudoephedrine 5 mg/240 mg Extended-Release Tablet and Clarinex-D® 24-Hour (Reference) Following a 5 mg/240 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Desloratadine and Pseudoephedrine Extended-release Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 50631
Record Dates: First submitted 2011-09-27; First posted 2012-01-10 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2006-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Desloratadine and pseudoephedrine; crossover
MeSH Terms: interventions — desloratadine; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Desloratadine and pseudoephedrine ER tablets 5/240 mg (Experimental): Desloratadine and pseudoephedrine ER tablets 5/240 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Desloratadine and pseudoephedrine
- Clarinex D 24-hour (Active Comparator): Clarinex D-24 of Schering Corporation Inc USA
  Interventions: Drug: Desloratadine and pseudoephedrine

INTERVENTIONS:
Drug: Desloratadine and pseudoephedrine — Desloratadine and pseudoephedrine 5/240 mg
  Other Names: Clarinex D-24

SUMMARY:
This is an open label, randomised, 2-way crossover, comparative bioequivalence study.

DETAILED DESCRIPTION:
The objective of this study was to compare the rate and extent of absorption of Dr. Reddy's Laboratories Ltd., India, desloratadine-pseudoephedrine and Schering Corporation, U.S.A.(Clarinex-D® 24-HOUR), desloratadine-pseudoephedrine, administered as a 1 x 5 mg/240 mg extended-release tablet under fed conditions. The treatment phases were separated by a washout period of 14 days. 44 subjects were dosed and were enrolled in the study; 43 of these enrolled subjects completed the study.

ELIGIBILITY:
Inclusion Criteria:

* Is the individual a healthy, normal adult man or woman who volunteers to participate?
* Is s/he within 18 to 45 years of age, inclusive?
* Is his/her BMI between 19 and 30 inclusive?
* Is she willing to avoid pregnancy by abstaining from sexual intercourse with a non-sterile male partner, or by the use one of the following methods: diaphragm + spermicide or condom + spermicide (at least 14 days before dosing), intra-uterine contraceptive device or hormonal contraceptives (at least 4 week prior to dosing) or has she been surgically sterile or post-menopausal at least six months prior to entering into the study?
* Is s/he considered reliable and capable of understanding his/her responsibility and role in the study?
* Has s/he provided written informed consent?

Exclusion Criteria:

* Does the individual have a history or allergy or hypersensitivity to desloratadine or pseudoephedrine, milk or eggs?
* Does s/he have clinically significant laboratory abnormalities that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Does s/he have significant history or clinical evidence of auto-immune, cardiovascular, gastrointestinal, hematological, hematopoietic, hepatic, neurological, ongoing infection, pancreatic, or renal disease that would interfere with the conduct or interpretation of the study or jeopardize his/her safety?
* Is she nursing?
* Does s/he have serious psychological illness?
* Does s/he have significant history (within the past year) or clinical evidence of alcohol or drug abuse?
* Does s/he have a positive urine drug screen or a positive HIV-I, or hepatitis B or C screen, or a positive pregnancy test?
* Is s/he unable to refrain from the use of alcohol or xanthine-containing foods or beverages during periods beginning 48 hours prior to study drug administration and ending when the last blood sample has been taken in each study period?
* Has s/he used any prescription drug, other than hormonal contraceptives, during the 14 day period prior to study initiation, or any OTC drug during the 72 hour period preceding study initiation?
* Is s/he unable to refrain from the use of all concomitant medications, other than hormonal contraceptives, during the study?
* Has s/he donated or lost blood or participated in a clinical study which involved the withdrawal of a large volume of blood (480 mL or more), during the six week period preceding study initiation?
* Has s/he donated plasma during the two week period preceding study initiation?
* Has s/he received an investigational drug during the 30 day period preceding study initiated?
* Has s/he used any tobacco products in the 3 months preceding drug administration?

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2006-04; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Area under curve(AUC) | Pre-dose 0.5,1,1.5,2,2.5,3,3.5,4,4.5,5,6,7,8,9,10,12,24,36,48,72,96,120 and 144 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Antonio R Pizarro, MD, Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Ft Myers Inc, Broadway, Florida, United States